CLINICAL TRIAL: NCT01132092
Title: The Normal Standard of Brainstem Auditory Evoked Potential in Adults Using a New Device
Status: Completed | Type: Observational
Sponsor: Universidade Estadual de Ciências da Saúde de Alagoas (Other)
Other Study IDs: UNCISAL-IS-001
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Normal Hearing (76 Subjects); Subjects With Hearing Loss (15 Subjects)
Keywords: Evoked Potentials, Adult, Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Normal hearing (experimental 1): 76 Normal hearing subjects, male and female, adults, , evaluated by new device
- Normal hearing (experimental 2): 15 Normal hearing subjects, male and female, adults, , evaluated by new device
- Hearing loss (experimental 3): 15 hearing loss subjects, male and female, adults, evaluated by new device
- Gold standard 1: 15 Normal hearing subjects, male and female, adults, evaluated by gold standard device
- Gold Standard 2: 15 hearing loss subjects, male and female, adults, evaluated by gold standard device

SUMMARY:
There are no differences between the exams made with the new device,that evaluates the hearing, and the device gold standard, that is widely used in clinics and hospitals.

ELIGIBILITY:
Inclusion Criteria:

* hearing thresholds less than 25 dB at all frequencies of pure tone audiometry, with differences between the ears, by frequency, or less than 10 dB.
* The group with bilateral sensorineural hearing loss was made up of adults with hearing thresholds changed from 25 to 60 dB HL for the frequencies 2000-8000 Hz for pure tone audiometry.

Exclusion Criteria:

-

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults Normal hearing subjects and hearing loss Subjects
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual de Ciências da Saúde de Alagoas, Maceió, Alagoas, Brazil